CLINICAL TRIAL: NCT01201473
Title: CONDOR Impact of Dental Practice-Based Research Network (PIRG)
Brief Title: CONDOR Impact of Dental Practice-Based Research Network
Acronym: CONDOR PIRG
Status: Completed | Type: Observational
Sponsor: Dental Practice-Based Research Network (Network)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); HealthPartners Institute (Other); Kaiser Permanente (Other); Permanente Dental Associates Group, Oregon (Other)
Responsible Party: Gregg H. Gilbert, DDS, MBA, Study Chair, The University of Alabama at Birmingham
Other Study IDs: 126171; U01DE016747 (NIH)
Record Dates: First submitted 2010-09-13; First posted 2010-09-14 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Behavior Changes
Keywords: effect of participation; effect of association

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Measure impact of research participation

SUMMARY:
The purpose of this study was to study the use of a Core Questionnaire that included several questions from each PBRN (DPBRN, PEARL, PRECEDENT - collectively know as CONDOR) that had been extracted from questionnaires previously administered as part of their initial research program activities. This protocol was the first administration of this core questionnaire with the purpose of assessing dental practice changes that may have occured since the earlier administration of the individual questions with the separate networks.It also collected baseline data for others.

DETAILED DESCRIPTION:
The three dental PBRNs had a unique opportunity to measure the impact of research participation on potential changes in practice base of the research protocol. We were able to examine the effect of participation in research in general to the acceptance of research findings from other studies and the effect of association with but not participation in a research network.

ELIGIBILITY:
Inclusion Criteria:

* DPBRN dentists and hygienists who had completed a DPBRN Enrollment questionnaire and for whom DPBRN had a current active address and who were currently licensed to practice
* reported on the Enrollment Questionnaire they were a general dentist, pediatric dentist, or dental hygienist, or reported doing at least some restorative dentistry procedures
* practiced in one of the five DPBRN regions (AL/MS, FL/GA, MN< PDA, or SK)

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The questionnaire was administered to all DPBRN practitioner-investigators (including both dentists and hygienists) 22 years of age or older.
Sampling Method: Non-Probability Sample
Enrollment: 687 (Actual)
Dates: Start 2009-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregg H Gilbert, DDS, MBA, Study Chair — The University of Alabama at Birmingham
Locations (7):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Florida College of Dentistry, Gainesville, Florida
  - Health Partners Dental Group, Minneapolis, Minnesota
  - Health Partners Research Foundation, Minneapolis, Minnesota
  - Kaiser Permanente Center for Health Research, Portland, Oregon
  - Permanente Denrtal Associates, Portland, Oregon
- University of Copenhagen Royal Dental College, Copenhagen, Denmark

REFERENCES:
- See also: Dental Practice-Based Research Network — http://DPBRN.org
- See also: Dental Practice-Based Research Network — http://DentalPBRN.org